CLINICAL TRIAL: NCT00876733
Title: Non-Interventional Observational Study With Viramune Plus ARV in HIV Infected Patients
Brief Title: Non-Interventional Observational Study With Viramune Plus Antiretroviral in HIV Infected Patients
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1100.1524
Record Dates: First submitted 2009-03-20; First posted 2009-04-07 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- HIV treatment

SUMMARY:
This observational study is supposed to assess (under conditions of clinical practice in daily routine) whether treatment with Viramune (nevirapine) in combination with ARV, e.g. Combivir (Zidovudine and Lamivudine), Kivexa (Abacavir and Lamivudine) or Truvada (tenofovir and emtricitabine) will durably suppress viral load below the limit of detection or will maintain suppression of viral replication (HIV-RNA below limit of detection) achieved under previous anti-retroviral combination therapy after switch to combination treatment of Viramune (nevirapine) and ARV, e.g. Combivir (Zidovudine and Lamivudine), Kivexa (Abacavir and Lamivudine) or Truvada (tenofovir and emtricitabine).

ELIGIBILITY:
Inclusion criteria:

* male and female
* 18 years or older
* written informed consent
* The inclusion criteria for treatment with Viramune plus other antiretroviral combination drugs are to be based on the current information for healthcare professionals / SmPC

Exclusion criteria:

* Pregnant patients
* The exclusion criteria for the treatment of Viramune plus other antiretroviral combination drugs are to be based on the current SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients
Sampling Method: Non-Probability Sample
Enrollment: 605 (Actual)
Dates: Start 2009-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (66):
- Germany (66):
  - Boehringer Ingelheim Investigational Site 14, Aachen
  - Boehringer Ingelheim Investigational Site 12, Berlin
  - Boehringer Ingelheim Investigational Site 13, Berlin
  - Boehringer Ingelheim Investigational Site 15, Berlin
  - Boehringer Ingelheim Investigational Site 19, Berlin
  - Boehringer Ingelheim Investigational Site 21, Berlin
  - Boehringer Ingelheim Investigational Site 23, Berlin
  - Boehringer Ingelheim Investigational Site 24, Berlin
  - Boehringer Ingelheim Investigational Site 28, Berlin
  - Boehringer Ingelheim Investigational Site 30, Berlin
  - Boehringer Ingelheim Investigational Site 31, Berlin
  - Boehringer Ingelheim Investigational Site 34, Berlin
  - Boehringer Ingelheim Investigational Site 38, Berlin
  - Boehringer Ingelheim Investigational Site 41, Berlin
  - Boehringer Ingelheim Investigational Site 54, Berlin
  - Boehringer Ingelheim Investigational Site 60, Berlin
  - Boehringer Ingelheim Investigational Site 63, Berlin
  - Boehringer Ingelheim Investigational Site 8, Berlin
  - Boehringer Ingelheim Investigational Site 58, Bochum
  - Boehringer Ingelheim Investigational Site 50, Chemnitz
  - Boehringer Ingelheim Investigational Site 53, Cologne
  - Boehringer Ingelheim Investigational Site 61, Cologne
  - Boehringer Ingelheim Investigational Site 48, Dortmund
  - Boehringer Ingelheim Investigational Site 27, Duisburg
  - Boehringer Ingelheim Investigational Site 49, Düsseldorf
  - Boehringer Ingelheim Investigational Site 62, Düsseldorf
  - Boehringer Ingelheim Investigational Site 9, Düsseldorf
  - Boehringer Ingelheim Investigational Site 32, Frankfurt
  - Boehringer Ingelheim Investigational Site 59, Frankfurt
  - Boehringer Ingelheim Investigational Site 65, Frankfurt
  - Boehringer Ingelheim Investigational Site 57, Freiburg im Breisgau
  - Boehringer Ingelheim Investigational Site 56, Fürth
  - Boehringer Ingelheim Investigational Site 29, Giessen
  - Boehringer Ingelheim Investigational Site 33, Hamburg
  - Boehringer Ingelheim Investigational Site 42, Hamburg
  - Boehringer Ingelheim Investigational Site 47, Hamburg
  - Boehringer Ingelheim Investigational Site 51, Hamburg
  - Boehringer Ingelheim Investigational Site 40, Hanover
  - Boehringer Ingelheim Investigational Site 43, Hanover
  - Boehringer Ingelheim Investigational Site 46, Hanover
  - Boehringer Ingelheim Investigational Site 6, Karlsruhe
  - Boehringer Ingelheim Investigational Site 25, Koblenz
  - Boehringer Ingelheim Investigational Site 37, Krefeld
  - Boehringer Ingelheim Investigational Site 11, Leipzig
  - Boehringer Ingelheim Investigational Site 52, Mainz
  - Boehringer Ingelheim Investigational Site 18, München
  - Boehringer Ingelheim Investigational Site 20, München
  - Boehringer Ingelheim Investigational Site 22, München
  - Boehringer Ingelheim Investigational Site 26, München
  - Boehringer Ingelheim Investigational Site 35, München
  - Boehringer Ingelheim Investigational Site 5, München
  - Boehringer Ingelheim Investigational Site 16, Münster
  - Boehringer Ingelheim Investigational Site 17, Münster
  - Boehringer Ingelheim Investigational Site 39, Münster
  - Boehringer Ingelheim Investigational Site 55, Münster
  - Boehringer Ingelheim Investigational Site 10, Neuss
  - Boehringer Ingelheim Investigational Site 36, Oldenburg
  - Boehringer Ingelheim Investigational Site 64, Osnabrück
  - Boehringer Ingelheim Investigational Site 7, Pforzheim
  - Boehringer Ingelheim Investigational Site 66, Potsdam
  - Boehringer Ingelheim Investigational Site 1, Stuttgart
  - Boehringer Ingelheim Investigational Site 3, Stuttgart
  - Boehringer Ingelheim Investigational Site 4, Stuttgart
  - Boehringer Ingelheim Investigational Site 45, Troisdorf
  - Boehringer Ingelheim Investigational Site 2, Wiesbaden
  - Boehringer Ingelheim Investigational Site 44, Wuppertal

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment-naive Patients: Patients who were not pretreated with HIV therapy.
- Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL: Patients switching from a virologically effective treatment regimen (i.e. due to intolerance), with a viral load ≤ 50 copies/mL.
- Pretreated Patients, Baseline Viral Load > 50 Copies/mL: Patients switching from a virologically ineffective treatment regimen, viral load >50 copies/mL.
- Patients With Baseline Viral Load Not Documented: Patients who could not be assigned to one of the three subgroups and had no documented viral load value.
Period: Overall Study
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Started | 288 | 203 | 93 | 21
Completed | 197 | 161 | 63 | 14
Not Completed | 91 | 42 | 30 | 7
Not completed — Adverse Event | 34 | 20 | 10 | 3
Not completed — Lack of Efficacy | 17 | 9 | 10 | 1
Not completed — Lost to Follow-up | 26 | 10 | 3 | 2
Not completed — Data not available | 14 | 3 | 7 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): This patient set includes all HIV-1 infected patients who were dispensed Viramune® and were documented to have taken at least one dose of Viramune®and of a antiretroviral combination partner.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented | Total
Number analyzed (Participants) | 288 | 203 | 93 | 21 | 605
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (9.9) | 43.8 (9.6) | 40.9 (9.4) | 43.6 (7.8) | 41.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 6 | 0 | 67
  Male | 256 | 174 | 87 | 21 | 538

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AE) and All Serious AEs
Description: Number of participants with Treatment Emergent Adverse Events (AE) and All Serious AEs
Time Frame: 36 months
Population: Patients from Full Analysis Set (FAS): This patient set includes all patients in the treated set who have analysable data in at least one efficacy endpoint.
Measure: Number; unit: participants
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 288 | 203 | 93 | 21
participants
  Patients with any AE | 168 | 110 | 51 | 10
  Patients with serious AEs | 17 | 12 | 5 | 0

2. Secondary Outcome: Changes in the Viral Load After 12 Months From Baseline.
Description: The change in the log10 viral load from baseline after 12 months was calculated by subtracting the baseline value from the value after 12 months. Therefore, a negative change represents a decrease in viral load.
Time Frame: Baseline and 12 months
Population: Patients from FAS with values for viral load at baseline and after 12 months.
Measure: Mean (Standard Deviation); unit: Log10 copies/ml
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 238 | 181 | 78 | 0
Log10 copies/ml | -3.3 (1.3) | -0.1 (0.8) | -1.9 (1.7) |

3. Secondary Outcome: Changes in the Viral Load After 36 Months From Baseline.
Description: The change in the log10 viral load from baseline after 36 months was calculated by subtracting the baseline value from the value after 36 months. Therefore, a negative change represents a decrease in viral load.
Time Frame: Baseline and 36 months
Population: Patients from FAS with values for viral load at baseline and after 36 months.
Measure: Mean (Standard Deviation); unit: Log10 copies/ml
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 231 | 185 | 74 | 0
Log10 copies/ml | -3.4 (1.4) | -0.2 (1.1) | -2.1 (1.8) |

4. Secondary Outcome: Changes in the Cluster of Differentiation 4 (CD4+) Cell Count After 12 Months From Baseline.
Description: The change in the CD4+ cell count from baseline after 12 months was calculated by subtracting the baseline value from the value after 12 months. Therefore, a positive change represents an increase in CD4+ cell count.
Time Frame: Baseline and 12 months
Population: Patients from FAS with values for CD4+ at baseline and after 12 months.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 238 | 178 | 76 | 2
cells/mm^3 | 188.7 (165.0) | 54.6 (145.3) | 82.8 (269.5) | 128.0 (223.4)

5. Secondary Outcome: Changes in the CD4+ Cell Count After 36 Months From Baseline.
Description: The change in the CD4+ cell count from baseline after 36 months was calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase in CD4+ cell count.
Time Frame: Baseline and 36 months
Population: Patients from FAS with values for CD4+ at baseline and after 36 months.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 230 | 181 | 72 | 2
cells/mm^3 | 223.7 (200.4) | 2.8 (221.3) | 116.0 (317.7) | 63.5 (152.0)

6. Secondary Outcome: Changes in the Laboratory Data (Total Cholesterol) After 12 Months From Baseline
Description: The changes in the laboratory data (Total Cholesterol) from baseline after 12 months were calculated by subtracting the baseline value from the value after 12 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 12 months
Population: Patients from TS with evaluable data for Total Cholesterol at baseline and at month 12.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 139 | 128 | 42 | 5
mg/dL | 25.2 (36.2) | -3.0 (43.2) | 15.8 (32.8) | 16.4 (9.7)

7. Secondary Outcome: Changes in the Laboratory Data (HDL Cholesterol) After 12 Months From Baseline
Description: The changes in the laboratory data ( High density protein (HDL) Cholesterol) from baseline after 12 months were calculated by subtracting the baseline value from the value after 12 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 12 months
Population: Patients from TS with evaluable data for HDL Cholesterol at baseline and at month 12.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 95 | 76 | 26 | 4
mg/dL | 12.7 (14.3) | 4.2 (15.0) | 10.9 (14.9) | -13.2 (29.1)

8. Secondary Outcome: Changes in the Laboratory Data (LDL Cholesterol) After 12 Months From Baseline
Description: The changes in the laboratory data ( Low density protein (LDL) Cholesterol) from baseline after 12 months were calculated by subtracting the baseline value from the value after 12 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 12 months
Population: Patients from TS with evaluable data for LDL Cholesterol at baseline and at month 12.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 95 | 75 | 25 | 4
mg/dL | 12.1 (29.6) | 2.4 (35.7) | 14.4 (30.5) | 13.6 (10.1)

9. Secondary Outcome: Changes in the Laboratory Data (Triglycerides) After 12 Months From Baseline
Description: The changes in the laboratory data (Triglycerides) from baseline after 12 months were calculated by subtracting the baseline value from the value after 12 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 12 months
Population: Patients from TS with evaluable data for Triglycerides at baseline and at month 12.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 139 | 130 | 38 | 5
mg/dL | 7.9 (106.7) | -61.6 (180.2) | -24.0 (78.9) | 16.3 (47.2)

10. Secondary Outcome: Changes in the Laboratory Data (Blood Glucose) After 12 Months From Baseline
Description: The changes in the laboratory data (Blood Glucose) from baseline after 12 months were calculated by subtracting the baseline value from the value after 12 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 12 months
Population: Patients from TS with evaluable data for Blood Glucose at baseline and at month 12.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 136 | 134 | 44 | 4
mg/dL | 0.2 (20.6) | -3.6 (16.9) | 0.3 (24.9) | -8.4 (9.2)

11. Secondary Outcome: Changes in the Laboratory Data (ALT) After 12 Months From Baseline
Description: The changes in the laboratory data (Alanine transaminase (ALT)) from baseline after 12 months were calculated by subtracting the baseline value from the value after 12 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 12 months
Population: Patients from TS with evaluable data for ALT at baseline and at month 12.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 175 | 152 | 49 | 7
U/L | 5.6 (20.5) | 10.2 (28.8) | 7.0 (28.4) | 9.7 (33.0)

12. Secondary Outcome: Changes in the Laboratory Data (AST) After 12 Months From Baseline
Description: The changes in the laboratory data (Aspartate transminase (AST)) from baseline after 12 months were calculated by subtracting the baseline value from the value after 12 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 12 months
Population: Patients from TS with evaluable data for AST at baseline and at month 12.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 173 | 146 | 48 | 7
U/L | 1.7 (19.1) | 4.4 (24.7) | 3.0 (20.9) | 8.3 (32.4)

13. Secondary Outcome: Changes in the Laboratory Data (Gamma GT) After 12 Months From Baseline
Description: The changes in the laboratory data (Gamma glutamyl transferase (Gamma GT)) from baseline after 12 months were calculated by subtracting the baseline value from the value after 12 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 12 months
Population: Patients from TS with evaluable data for Gamma GT at baseline and at month 12.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 175 | 152 | 49 | 7
U/L | 32.9 (72.4) | 25.4 (57.7) | 23.7 (62.3) | 9.1 (42.6)

14. Secondary Outcome: Changes in the Laboratory Data (Creatinine) After 12 Months From Baseline
Description: The changes in the laboratory data (Creatinine) from baseline after 12 months were calculated by subtracting the baseline value from the value after 12 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 12 months
Population: Patients from TS with evaluable data for Creatinine at baseline and at month 12.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 176 | 152 | 47 | 7
mg/dL | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.2)

15. Secondary Outcome: Changes in the Laboratory Data (Haemoglobin) After 12 Months From Baseline
Description: The changes in the laboratory data (Haemoglobin) from baseline after 12 months were calculated by subtracting the baseline value from the value after 12 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 12 months
Population: Patients from TS with evaluable data for Haemoglobin at baseline and at month 12.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 177 | 147 | 45 | 7
g/dL | 0.6 (1.1) | 0.3 (1.2) | 0.3 (0.9) | 0.5 (1.1)

16. Secondary Outcome: Changes in the Laboratory Data (Total Cholesterol) After 36 Months From Baseline
Description: The changes in the laboratory data (Total Cholesterol) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for Total Cholesterol at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 82 | 66 | 25 | 2
mg/dL | 24.1 (39.0) | 2.0 (44.4) | 24.2 (42.4) | 41.1 (12.9)

17. Secondary Outcome: Changes in the Laboratory Data (HDL Cholesterol) After 36 Months From Baseline
Description: The changes in the laboratory data ( High density protein (HDL) Cholesterol) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for HDL Cholesterol at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 53 | 42 | 15 | 2
mg/dL | 11.0 (21.4) | 4.4 (20.7) | 11.1 (11.9) | -19.6 (38.7)

18. Secondary Outcome: Changes in the Laboratory Data (LDL Cholesterol) After 36 Months From Baseline
Description: The changes in the laboratory data ( Low density protein (LDL) Cholesterol) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for LDL Cholesterol at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 53 | 40 | 15 | 2
mg/dL | 12.4 (25.8) | 15.8 (38.1) | 23.8 (44.7) | 22.7 (27.9)

19. Secondary Outcome: Changes in the Laboratory Data (Triglycerides) After 36 Months From Baseline
Description: The changes in the laboratory data (Triglycerides) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for Triglycerides at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 83 | 67 | 25 | 1
mg/dL | -3.4 (91.3) | -73.7 (252.6) | -17.2 (98.0) | 34.2

20. Secondary Outcome: Changes in the Laboratory Data (Blood Glucose) After 36 Months From Baseline
Description: The changes in the laboratory data (Blood Glucose) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for Blood Glucose at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 78 | 71 | 23 | 1
mg/dL | 1.6 (27.2) | 0.0 (19.9) | 0.7 (36.4) | -7.2

21. Secondary Outcome: Changes in the Laboratory Data (ALT) After 36 Months From Baseline
Description: The changes in the laboratory data (Alanine transaminase (ALT)) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for ALT at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 103 | 76 | 30 | 3
U/L | 16.2 (107.1) | 4.0 (33.7) | 11.8 (27.7) | 5.2 (26.1)

22. Secondary Outcome: Changes in the Laboratory Data (AST) After 36 Months From Baseline
Description: The changes in the laboratory data (Aspartate transminase (AST)) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for AST at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 100 | 75 | 29 | 3
U/L | 7.3 (75.3) | 0.1 (24.6) | 5.5 (27.1) | -2.7 (19.6)

23. Secondary Outcome: Changes in the Laboratory Data (Gamma GT) After 36 Months From Baseline
Description: The changes in the laboratory data (Gamma glutamyl transferase (Gamma GT)) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for Gamma GT at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 104 | 76 | 30 | 3
U/L | 52.3 (102.5) | 45.0 (112.6) | 50.3 (50.3) | 12.9 (48.1)

24. Secondary Outcome: Changes in the Laboratory Data (Creatinine) After 36 Months From Baseline
Description: The changes in the laboratory data (Creatinine) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for Creatinine at baseline and at month 12.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 103 | 74 | 30 | 3
mg/dL | 0.0 (0.2) | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1)

25. Secondary Outcome: Changes in the Laboratory Data (Haemoglobin) After 36 Months From Baseline
Description: The changes in the laboratory data (Haemoglobin) from baseline after 36 months were calculated by subtracting the baseline value from the value after 36 months. Therefore, a positive change represents an increase, a negative change represents a decrease in the data.
Time Frame: Baseline and 36 months
Population: Patients from TS with evaluable data for Haemoglobin at baseline and at month 36.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Number analyzed (Participants) | 103 | 73 | 30 | 3
g/dL | 0.7 (0.9) | 0.2 (1.2) | 0.5 (1.4) | -0.1 (1.6)

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Treatment-naive Patients | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL | Pretreated Patients, Baseline Viral Load > 50 Copies/mL | Patients With Baseline Viral Load Not Documented
Serious Adverse Events (participants affected / at risk) | 17/288 | 12/203 | 5/93 | 0/21
Other Adverse Events (participants affected / at risk) | 51/288 | 33/203 | 22/93 | 3/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-naive Patients (N=288) | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL (N=203) | Pretreated Patients, Baseline Viral Load > 50 Copies/mL (N=93) | Patients With Baseline Viral Load Not Documented (N=21)
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Device occlusion (General disorders) | 0 | 1 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 0 | 0
Tenderness (General disorders) | 1 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Acute hepatitis C (Infections and infestations) | 1 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 1 | 0
Meningoencephalitis herpetic (Infections and infestations) | 0 | 0 | 1 | 0
Myelitis (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Biopsy (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hypopharyngeal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 2 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Somatoform disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bursa removal (Surgical and medical procedures) | 0 | 0 | 1 | 0
Laparoscopic surgery (Surgical and medical procedures) | 0 | 1 | 0 | 0
Laser therapy (Surgical and medical procedures) | 1 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment-naive Patients (N=288) | Pretreated Patients, Baseline Viral Load ≤ 50 Copies/mL (N=203) | Pretreated Patients, Baseline Viral Load > 50 Copies/mL (N=93) | Patients With Baseline Viral Load Not Documented (N=21)
Diarrhoea (Gastrointestinal disorders) | 16 | 14 | 7 | 2
Bronchitis (Infections and infestations) | 14 | 21 | 9 | 1
Nasopharyngitis (Infections and infestations) | 30 | 13 | 15 | 1
Upper respiratory tract infection (Infections and infestations) | 15 | 3 | 3 | 0
Transaminase increased (Investigations) | 16 | 3 | 2 | 0
Hypertension (Vascular disorders) | 8 | 6 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.